CLINICAL TRIAL: NCT04446689
Title: Biofeedback Efects on Stress, Anxiety, and Quality of Professional Life on Nursing Staff of an University Hospital
Brief Title: Biofeedback Effects on Nursing Personal at an University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-06-45
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Stress (Psychology); Biofeedback, Psychology
Keywords: nursing staff
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Active Comparator): The intervention group will develop an activity with self-monitoring called Cardiovascular Biofeedback or Cardiac Frequency Variability (CFV). This intervention will be measured by the Software Emwave Pro Plus during 4 weeks, which send out a sign captured by a non-invasive sensor such as an ear lobe fixed photoplethysmograph. This photoplethysmograph verifies blood flow alterations through an optical method. Cardiac frequency oscillations may be estimated both by the quantity of blood infrared lights absorbed or reflected, and by variations in blood volume and pressure. Captured physiological signs will be recorded during ten minutes by the Software Emwave Pro Plus®, which is adapted to biofeedback training.
  Interventions: Behavioral: Biofeedback
- activity without self monitoring (No Intervention): The placebo group will develop an activity without self monitoring. In order to keep blindness between the groups the activities will be processed by an electronic device - the on line app Jigsaw Puzzles. This app consists of a puzzle with different levels of difficulties, and is played in a tablet.
  Each participant will be performing in the study during four weeks, with two encounters each week (total: four weeks). While the participant will be performing its activity he/she will be monitored by the researchers through CFV (Cardiac Frequency Variability) - with no visualization of the computer monitor.
  The control group will answer the research protocol in two moments (D1 and D8), to evaluate

INTERVENTIONS:
Behavioral: Biofeedback — This intervention will be measured by the Software Emwave Pro Plus during 4 weeks, which send out a sign captured by a non-invasive sensor such as an ear lobe fixed photoplethysmograph.
  Arms: Biofeedback

SUMMARY:
Randomized Clinical Trial comparing two groups: placebo group without self-monitoring of heart rate variability (HRV) and biofeedback intervention that includes self-monitoring of HRV

DETAILED DESCRIPTION:
Its main objective is to evaluate the effects of Biofeedback intervention on the stress, and anxiety levels, as well as the quality of professional life, and their coping mechanisms, of a nursing staff from de Hospital de Clínicas de Porto Alegre. The research will have two phases, first to select the nursing staff sample, and then to apply and evaluate the intervention. From 2.219 individuals will be randomly drawn a sample of 272 participants. All will respond a questionnaire (Vasconcelos Symptoms and Stress List) in order to obtain a general level of stress score greater than 1 (inclusion criteria to enter the RCT). The 272 group will be randomly split in two groups (136 subjects each) to compare the intervention vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff
* Both sexes
* Working activities
* Admitted in the last 90 days
* Presenting a level stress greater then 1

Exclusion Criteria:

* Pregnant and breast feeding professionals
* Those away from work a long time, and or returning from vacations in the last 15 days. ----Participants with any kind of cardiac pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Stress | 4 weeks
  Stress evaluation will be measured by the 23 items Work Stress Scale (WST), likert scale with each item corresponding to a stressor and the reaction the subject has to it. Scores vary from 23 to 111 points, with good reliability (COM µ = 0,91). Results were obtained by the items media sum, considering occupational stress as low (values between 1 and 2), moderate (2,01 to 2,99), or high (3 to 5).

CONTACTS AND LOCATIONS:
Overall Officials: Sônia Souza, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil